CLINICAL TRIAL: NCT01767051
Title: Children Follow-up of PCOS Women.Cardiovascular Health in Offspring of PCOS Mothers
Brief Title: Children Follow-up of PCOS Women
Acronym: CHOPS
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Bart CJM Fauser, Professor of Reproductive Medicine, UMC Utrecht
Other Study IDs: CHOPS METC 12/308
Record Dates: First submitted 2013-01-08; First posted 2013-01-11 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Cardiovascular Health; Metabolic Health; Pulmonary Health
Keywords: PCOS; Children; Cardiovascular; Follow-up

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — saliva, serum, plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Children born from mothers who are diagnosed with PCOS: Children at the age of 2.5-4 years or at the age of 6-8 years born from mothers who are diagnosed with PCOS at the University Medical Centre in Utrecht (UMCU) in the period 2004-2012 (n=891) will be asked to participate. Children who were born before the diagnosed PCOS of their mothers at the UMCU will be asked to participate too. All mothers have been diagnosed with PCOS according to standardised extensive diagnostic work-up and have given informed consent to be approached for future research purposes.
- Children who participated in the WHISTLER study: Children who participated in the WHISTLER 3 (11-163) and WHISTLER/Cardio study (10-194) in 2002-2012. The children were born from mothers with a regular cycle prior to conception who conceived naturally. The children were examined at the age of 2.5-4 years or at the age of 7-8 years. The data of the WHISTLER 3 and WHISTLER/Cardio study have already been collected.

SUMMARY:
Polycystic ovary syndrome (PCOS) is a complex and frequent disorder with a heterogeneous clinical presentation varying throughout life, from birth up to post-menopause. Although mostly known for its reproductive consequences, PCOS is associated with metabolic abnormalities related to insulin resistance and obesity. Children born from PCOS mothers are considered to be at risk for early insulin resistance, leading to development of PCOS and metabolic abnormalities in childhood and adolescence. Obesity and insulin resistance are considered as states of low- and pro-inflammation associated with endothelial dysfunction. In addition, it has been shown that endothelial dysfunction develops from the first decade of life in response to genetic and environmental risk factors. Therefore, offspring of women with PCOS may be at increased risk for vascular disease later in life. Moreover, some evidence suggests that early life respiratory disease also contributes to later life cardiovascular consequences. The number of studies on offspring of PCOS mothers is low and a systematic follow up of children born form PCOS mothers has not been performed yet. the investigators propose a systematic evaluation of cardiometabolic and pulmonary health characteristics of children (aged 2,5-8 years) born from mothers diagnosed with PCOS. A saliva sample will be performed to determine the biochemical androgenic status of the children. Mothers of these children have undergone standardized phenotyping prior to conception; the investigators will therefore be able to correlate the metabolic status of the mother around the time of conception and the cardiometabolic and pulmonary health of their offspring.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Children
* Children participating in WHISTLER study or children of PCOS mothers
* Aged 2.5-4 years or 6-8 years

Exclusion Criteria:

* Language barrier
* Children with a history of a heart defect
* Children with a respiratory infection or respiratory infection two weeks previous to the visit are asked to reschedule the appointment.
* Residency outside the Netherlands
* Diabetes Mellitus type I
* Unresolved medical conditions

Ages: 30 Months to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Cases Children born from mothers who are diagnosed with PCOS at the UMCU will be asked to participate. Children who were born before the diagnosed PCOS of their mothers at the UMCU will be asked to participate too. All mothers have been diagnosed with PCOS according to standardised extensive diagnostic work-up and have given informed consent to be approached for future research purposes.
  Controls Children who participated in the WHISTLER study (protocol number 10-194) in . The children were born from mothers with a regular cycle prior to conception and who conceived naturally. The children were examined at the age of 2.5-4 years or at the age of 6-8 years. The data of the WHISTLER 3 and WHISTLER/Cardio study have already been collected.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pulse wave velocity (age 2.5-4 years) | 12 months
  The pulse wave velocity will be measured twice using the Arteriograph at the right arm. This measurement will start by performing a blood pressure measurement at the first phase. In the second phase the pulse wave recording for pulse waveform analysis is performed. First the device will inflate back to the measured diastolic value and register the pulse waves and second, the device inflates further to the suprasystolic value (to the measured systolic value +35 mmHg), occluding the brachial artery completely in this way and registers the pulse waves.
Echocardiography (age 2.5-4 years) | 12 months
  Echocardiography will be performed in a supine position. Three ECG electrodes will be attached on the skin. The child can watch a movie during the measurements. Using M-mode and Tissue Doppler Echocardiography several measurements of the systolic and diastolic function of the right and left ventricle will be performed.
Anthropometry (both age categories) | 12 months
  Body height and weight will be measured to the nearest 0.1 cm and 0.1 kg respectively without wearing shoes. Distance between the jugular fossa and symphysis will be measured (needed for calculation of pulse wave velocity). Waist circumference will be measured twice at the bare skin using a non-elastic measuring tape, between the superior iliac anterior spine and the lowest rib in a horizontal line, at the end of a normal expiration. Hip circumference will be measured twice over light clothing at the most posterior point of the buttocks. Thoracic circumference will be measured at the end of the expiration and signs of respiratory disease will be noted.
Carotid intima media thickness (age 6-8 years) | 12 months
  The carotid IMT will be determined by using ultrasound based on the gold standard Wall Track System (Art.lab System, Esaote and the Cardiovascular Research Institute Maastricht).
Fat mass determination (6-8 years) | 12 months
  The intra-abdominal fat will be assessed by ultrasound by determination of the distance between the posterior side of the linea alba and the anterior vertebrae. The subcutaneous fat will be determined by measuring the distance between the anterior side of the linea alba and the skin. Both fat compartments will be assessed longitudinally.
Blood sample (6-8 years) | 12 months
  The venous puncture will be performed for the collection of the blood sample by using a butterfly needle, since this needle is smaller than the needles commonly used for venous puncture (vacutainer system) and will therefore reduce the pain of the venous puncture for the children. The venipuncture will be performed in a vein in the cubital fossa. Two different tubes of blood will be drawn, one sodium-heparin and one lithium-heparin tube, with in total a maximum of 19 cc blood. Prior to the venous puncture, a local anaesthetic, xylocaine spray, will be used at the location of the puncture.

SECONDARY OUTCOMES:
Airway resistance (both age categories) | 12 months
  Measurements of the airway resistance will be measured with the MicroRint using the interrupter technique according to standardized criteria. The child breathes passively through a mouthpiece. A rapidly occluding valve automatically interrupts the airflow for a period so brief as to be imperceptible to the patient. The airway resistance will automatically be computed.
Saliva sample (both age categories) | 12 months
  Saliva will be collected unstimulated by spittinh in a paper cup or with a Salimetrics children's swab. The saliva will be stored in a freezer (-80 degrees)
Flow-volume measurements | 12 months
  Flow-volume measurements will be performed by using spirometry.
Inflammatory markers in exhailed air | 12 months
  Nitric Oxide levels will be measured in exhaled air

CONTACTS AND LOCATIONS:
Locations (1):
- University medical Center Utrecht, Utrecht, Utrecht, Netherlands